CLINICAL TRIAL: NCT04903405
Title: Immune Function Monitoring and Immunotherapy in Sepsis: a Cross-sectional Survey in China
Brief Title: Immune Function Monitoring and Immunotherapy in Sepsis
Acronym: IMITS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Wu Jianfeng, chief physician, Sun Yat-sen University
Other Study IDs: IMITS
Record Dates: First submitted 2021-05-23; First posted 2021-05-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Sepsis; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sepsis
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention is involved in this study

SUMMARY:
At present, the clinical studies of various anti-inflammatory drugs and immune-enhancing drugs show that immunotherapy will bring new hope for the treatment of sepsis. In order to further understand the current status of immunotherapy in China, this study aims to understand the current status and standardization of the use of sepsis immunosurveillance and immunotherapy in hospitals through a cross-sectional survey.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sepsis or septic shock according to Sepsis 3.0

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient was diagnosed with sepsis or septic shock according to Sepsis 3.0
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | 28 days

SECONDARY OUTCOMES:
Percentage of sepsis patients receiving immune function monitoring | 28 days
Percentage of sepsis patients receiving immunotherapy | 28 days

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pei F, Zhang GR, Zhou LX, Liu JY, Ma G, Kou QY, He ZJ, Chen MY, Nie Y, Wu JF, Guan XD; China Critical Care Immunotherapy Research Group. Early Immunoparalysis Was Associated with Poor Prognosis in Elderly Patients with Sepsis: Secondary Analysis of the ETASS Study. Infect Drug Resist. 2020 Jun 30;13:2053-2061. doi: 10.2147/IDR.S246513. eCollection 2020. PMID 32636658
- [Background] Wu J, Zhou L, Liu J, Ma G, Kou Q, He Z, Chen J, Ou-Yang B, Chen M, Li Y, Wu X, Gu B, Chen L, Zou Z, Qiang X, Chen Y, Lin A, Zhang G, Guan X. The efficacy of thymosin alpha 1 for severe sepsis (ETASS): a multicenter, single-blind, randomized and controlled trial. Crit Care. 2013 Jan 17;17(1):R8. doi: 10.1186/cc11932. PMID 23327199
- [Background] Wu JF, Ma J, Chen J, Ou-Yang B, Chen MY, Li LF, Liu YJ, Lin AH, Guan XD. Changes of monocyte human leukocyte antigen-DR expression as a reliable predictor of mortality in severe sepsis. Crit Care. 2011;15(5):R220. doi: 10.1186/cc10457. Epub 2011 Sep 20. PMID 21933399